CLINICAL TRIAL: NCT01858792
Title: Efficacy and Safety of Belimumab in a Subgroup of Systemic Lupus Erythematosus (SLE) Patients With Higher Disease Activity (Anti-dsDNA Positive and Low Complement): A Pooled Analysis of the HGS1006-C1056 (BLISS-52) and HGS1006-C1057 (BLISS-76) Studies
Brief Title: A Pooled Analysis of the HGS1006-C1056 (BLISS-52) and HGS1006-C1057 (BLISS-76) Studies
Status: Completed | Type: Observational
Sponsor: Human Genome Sciences Inc., a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Other Study IDs: 115030
Record Dates: First submitted 2012-12-19; First posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Lupus Erythematosus, Discoid
MeSH Terms: conditions — Lupus Erythematosus, Discoid | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Baseline Health-Related Quality of Life (HRQOL): Quality of life assessment tools were similar across the treatment groups and indicated that there was impairment in quality of life of subjects in the Low C+anti-dsDNA Population
  Interventions: Drug: Belimumab 1 mg/kg; Drug: Belimumab 10 mg/kg; Other: Placebo
- SLE Medication Usage at Baseline: All subjects in the Low C+anti-dsDNA Population
  Interventions: Drug: Belimumab 1 mg/kg; Drug: Belimumab 10 mg/kg; Other: Placebo

INTERVENTIONS:
Drug: Belimumab 1 mg/kg — Belimumab 1 mg/kg IV plus standard therapy; belimumab 1 mg/kg administered on Days 0, 14, 28, and every 28 days thereafter through 72 weeks.
Drug: Belimumab 10 mg/kg — Belimumab 10 mg/kg IV plus standard therapy; belimumab 10 mg/kg administered on Days 0, 14, 28, and every 28 days thereafter through 72 weeks.
Other: Placebo — Placebo IV plus standard therapy; placebo administered on Days 0, 14, 28, and every 28 days thereafter through 72 weeks.

SUMMARY:
Efficacy and Safety of Belimumab in a Subgroup of Systemic Lupus Erythematosus (SLE) Patients with Higher Disease Activity (anti-dsDNA positive and low complement): A Pooled Analysis of the HGS1006-C1056 (BLISS-52) and HGS1006-C1057 (BLISS-76) Studies

DETAILED DESCRIPTION:
Studies C1056 and C1057 followed very similar protocols, were of nearly identical design, had common inclusion and exclusion criteria, and were conducted over the same time period. Nevertheless, given the heterogeneous presentation of SLE disease and the fact that the Phase III program was run globally, variation in the patient population, both within the studies (e.g., between different centres) and between the studies (analogous to differences between centres within the same study) should be expected.

Since it has been established that the conduct of the studies was effectively the same, it then must be determined whether the relative treatment effect is different in one study compared with the other study when evaluating whether two studies are similar enough to pool. Each of these Phase III studies achieved statistical significance for belimumab 10 mg/kg on the pre-specified primary endpoint of SRI response at Week 52; therefore, these nearly identical studies provide independent replication of results. While pooling is not necessary to establish the effectiveness of belimumab, it was considered appropriate in order to evaluate treatment effects in the high disease activity subgroup of interest, given that the individual studies were not designed to provide sufficient power to demonstrate effectiveness within subgroups. Thus, statistical evaluation pooling the studies and testing for a treatment-by-study interaction was undertaken. A significant treatment-by-study interaction would indicate that the relative treatment differences were statistically different in the two studies and pooling would not be justified. Conversely, the lack of a treatment-by-study interaction would indicate the studies resulted in a similar treatment response and pooling would be justified.

When the two Phase III studies were pooled for the SRI analysis, the treatment-by-study interaction was >0.5. Likewise, for the target population of high disease activity, the treatment-by-study interaction was >0.7 suggesting that the high disease activity subgroup may be more homogenous and therefore have a more similar treatment effect between the studies than the population as a whole.

Given these considerations, it is reasonable and valid to pool the two studies and allows better precision for evaluation of subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SLE by ACR criteria.
* Active SLE disease.
* Autoantibody-positive.
* On stable SLE treatment regimen.

Exclusion Criteria:

* Pregnant or nursing
* Have received treatment with any B cell targeted therapy.
* Have received treatment with a biological investigational agent in the past year.
* Have received IV cyclophosphamide within 180 days of Day 0.
* Have severe lupus kidney disease.
* Have active central nervous system (CNS) lupus.
* Have required management of acute or chronic infections within the past 60 days.
* Have current drug or alcohol abuse or dependence.
* Have a historically positive test or test positive at screening for HIV, hepatitis B, or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who were anti-dsDNA positive and had low C3 and/or C4 at baseline (Low C+anti-dsDNA Population) Subjects with baseline SELENA SLEDAI score >= 10 (SS >=10 Population)
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
SLE (systemic lupus erythematosus) Response Index (SRI) at Week 52 | Response rate by visit through Week 52 for the pooled studies and through Week 76 for Study C1056
  Composite endpoint resulting from the combination of three well-established tools for evaluating SLE disease activity which include an objective measure of the reduction in global disease activity for efficacy and two measures to ensure that the improvement in disease activity (score) is not offset by worsening of the subject's condition overall.

SECONDARY OUTCOMES:
The response rate by visit modified to exclude anti-dsDNA and complement items in the determination of a 4-point reduction in SELENA SLEDAI (Safety of Oestrogen in Lupus National Assessment Systemic Lupus Erythematosus Disease Activity Index). | By visit up to Week 52 for pooled studies.
The percent of subjects with no new BILAG A (British Isles Lupus Assessment Group) organ domain score or 2 new BILAG B organ domain scores | By visit up to Week 52 for pooled studies
Percent of subjects with greater than 4 point reduction from baseline in SELENA SLEDAI (Safety of Oestrogen in Lupus National Assessment Systemic Lupus Erythematosus Disease Activity Index) | By visit up to Week 52
Mean change in PGA (Physician's Global Assessment) | At Week 24, and by visit up to week 52 (population a only).
All Flares and Severe Flares will be assessed for population a | In periods of Weeks 0-52 and weeks 24-52
  Number of subjects experiencing a flare/severe flare (Weeks 0-52 and Weeks 24-52). Time to 1st flare/severe flare (Weeks 0-52 and Weeks 24-52.) Flares/Severe flares per subject year (Weeks 0-52).
All BILAG A (British Isles Lupus Assessment Group) Flares will be assessed for population a | In periods of Weeks 0-52 and Weeks 24-52
  Number of subjects experiencing a BILAG A flare (Weeks 0-52 and Weeks 24-52). Time to 1st BILAG A flare (Weeks 0-52 and Weeks 24-52). BILAG A flares per subject year (Weeks 0-52).
Percent of Subjects with Daily Prednisone Dose Reduced to ≤ 7.5 mg/day from > 7.5 mg/day at Baseline by Visit | For pooled studies through Week 52
Mean change in SF-36 (Short Form 36 Health Survey questionnaire) domains (population a only), Physical Component Summary (PCS) and Mental Component Summary MCS (population a only) | By visit up to Week 52
Mean change in FACIT (Functional Assessment of Chronic Illness Therapy) Fatigue Scale score | By visit up to Week 52
EQ-5D (EuroQol five dimension self-reported health state questionnaire) individual item score (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) | Change from baseline by visit up to Week 52
Improvement in each SELENA SLEDAI (Safety of Oestrogen in Lupus National Assessment Systemic Lupus Erythematosus Disease Activity Index) organ domain | At week 52
Percent of subjects with no worsening in PGA (Physician's Global Assessment) | By visit up to Week 52
Percent of Subjects with Daily Prednisone Dose Increased to > 7.5 mg/day from ≤7.5 mg/day at Baseline by Visit | For pooled studies through Week 52.
Percent of Subjects with Daily Prednisone Dose Reduced by ≥25% and to ≤ 7.5 mg/day from > 7.5 mg/day at Baseline by Visit | For pooled studies through Week 52
Time to first SELENA SLEDAI (Safety of Oestrogen in Lupus National Assessment Systemic Lupus Erythematosus Disease Activity Index) organ improvement by organ domain, among subjects with involvement at baseline | Over Weeks 0-52
Time to first BILAG organ improvement by organ domain, among subjects with involvement at baseline | Over Weeks 0-52
EQ-5D (EuroQol five dimension self-reported health state questionnaire) index score using value set for the UK | Change from baseline by visit up to Week 52
EQ-5D (EuroQol five dimension self-reported health state questionnaire) visual analogue scale (VAS) score using value set for the UK | Change from baseline by visit up to Week 52
The response rate calculated without allowable and prohibited medication rules applied (population a only). | By visit up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] van Vollenhoven RF, Petri MA, Cervera R, Roth DA, Ji BN, Kleoudis CS, Zhong ZJ, Freimuth W. Belimumab in the treatment of systemic lupus erythematosus: high disease activity predictors of response. Ann Rheum Dis. 2012 Aug;71(8):1343-9. doi: 10.1136/annrheumdis-2011-200937. Epub 2012 Feb 15. PMID 22337213